CLINICAL TRIAL: NCT00386893
Title: Influence of Escitalopram on Somatosensory Processing in Patients With Major Depression
Brief Title: Somatosensory Processing in Depression
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Principal Investigator, Oliver Pogarell, Investigator, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ESC_03082005; 2005-003752-35
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Magnetic Resonance Imaging

ARMS (1):
- Treatment as usual (Other): simultaneous EEG/fMRI
  Interventions: Procedure: simultaneous EEG/fMRI; Device: fMRI

INTERVENTIONS:
Procedure: simultaneous EEG/fMRI — fMRI/EEG recordings
Device: fMRI

SUMMARY:
Aim of this study is to investigate neuronal differences (EEG/evoked potentials; functional MRI) between patients with major depression and healthy controls concerning brain activity after acute pain as well as changes of pain related brain activity during treatment with escitalopram.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric in or outpatients with acute depressive episode
* Indication for pharmacological treatment

Exclusion Criteria:

* Acute suicidal tendency
* Neurological or severe somatic disorders
* Women during pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
changes in evoked potentials/functional MRI from baseline to week 4 | two assessments, at baseline and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Hegerl, MD, Principal Investigator — Department of Psychiatry, Ludwig-Maximilians-University; Oliver Pogarell, MD, Principal Investigator — Department of Psychiatry, Ludwig-Maximilians-University
Locations (1):
- Department of Psychiatry and Clin. Radiology, Ludwig-Maximilian-University, Munich, Bavaria, Germany